CLINICAL TRIAL: NCT05735782
Title: Association of Symptoms, Clinical and Biochemical Characteristics in Post COVID-19 Syndrome: a Case-control Study
Brief Title: Clinical and Biological Characterization of Post COVID-19 Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arturo Jauretche National University (Other)
Collaborators: Hospital El Cruce (Other); National University of Cuyo (Other); Universidad Nacional de La Plata (Other); University of Buenos Aires (Other)
Responsible Party: Principal Investigator, Laura Antonietti, Principal Investigator, Arturo Jauretche National University
Other Study IDs: PICTO-COVID-SECUELAS-00015
Record Dates: First submitted 2023-02-16; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Long COVID
Keywords: Post-Acute COVID-19 Syndrome; Long COVID; Post-COVID Conditions; Post Acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case-Control: Case group: Participants with persistent symptoms post-COVID-19 more than12 weeks after COVID-19 acute infection Control group: Participants without persistent symptoms after a COVID-19 acute infection.
  Interventions: Diagnostic Test: Clinical, mental health and psychosocial profile of Post-COVID-19 syndrome; Diagnostic Test: Diagnostic performance of echocardiographic and biological markers in Post-COVID-19 syndrome

INTERVENTIONS:
Diagnostic Test: Clinical, mental health and psychosocial profile of Post-COVID-19 syndrome — Evaluation of persistent symptoms of COVID-19 and its association with psychological, cognitive and social status in comparison to a healthy control group
Diagnostic Test: Diagnostic performance of echocardiographic and biological markers in Post-COVID-19 syndrome — Determine the inflammatory, immune profile and ventricular function in post-COVID-19 participants compared to a control group

SUMMARY:
The goal of this observational study is to describe the symptoms that persist for more than 12 weeks after the acute episode in participants who had COVID-19, and compare the functional, socioeconomic and occupational effects with a post-COVID-19 control group without persistent symptoms after the COVID-19 acute event.

The main questions it aims to answer are:

* What are the characteristics of symptoms that persist for more than 12 weeks in participants who have had COVID19 in the last year?
* What are the health-related quality of life and psychosocial effects in participants with persistent symptoms of COVID-19, compared to a post-COVID-19 control group without persistent symptoms after the acute episode of COVID-19?

DETAILED DESCRIPTION:
Two groups of cases and one group of controls will be included. A group of cases with persistent respiratory and/or cardiovascular symptoms (cardiorespiratory cases), and another group with persistent non-cardiorespiratory symptoms.

Participants who report at least two symptoms of intensity greater than or equal to severe will be classified as non-cardiorespiratory cases.

Controls will be participants with a history of confirmed SARS-CoV-2 infection, but without current or past persistent symptoms (ie, who resolved their symptoms during the acute episode or whose symptoms did not persist more than 4 weeks after onset).

Controls will be matched to cases by sex, age (with a margin of up to ±5 years), and time since diagnosis of the COVID-19 episode considered as the origin of post-COVID-19 symptoms in the cases (with a margin of of ±30 days).

The visit will include the application of the questionnaires for the evaluation of symptoms and quality of life associated with health, the clinical evaluation and the extraction of a blood sample.

The extraction of a blood sample will allow biochemical determinations, the complete blood count and vitamin D level to be carried out. Subsequently, an aliquot will be reserved for mechanistic evaluation (inflammatory markers, immunological and microRNA studies).

ELIGIBILITY:
Two groups of cases and one group of controls will be included. A group of cases with persistent respiratory and/or cardiovascular symptoms (cardiorespiratory cases), and another group with persistent non-cardiorespiratory symptoms. For participation in the study, people who meet the following inclusion criteria and none of the exclusion criteria will be considered.

Inclusion Criteria:

* Age equal to or greater than 18 years;
* Documented SARS-CoV-2 infection by PCR or antigen test;
* Ability to understand the objectives of the study;
* Acceptance to participate in the study and willingness to sign the informed consent.
* Permanent residence in Buenos Aires Metropolitan Area.

Exclusion Criteria:

* Women who report being pregnant, who are in the puerperium or lactation period at the time of the evaluation.
* People with known chronic debilitating conditions, defined as:

  i. heart failure, ii. symptomatic Coronary Heart Disease, iii. Diagnosis of cancer in the last 5 years iv. symptomatic anemia, v. chronic obstructive pulmonary disease or greater than moderate asthma, vi. heart valve disease more than mild, vii. cognitive impairment prior to the diagnosis of COVID-19, viii. diagnosis of schizophrenia or depression, ix. any other condition that, at the discretion of the treating professional or the research team, may explain or justify the aforementioned symptoms.
* Participants who are undergoing an acute pathology or who have undergone it in the last 4 weeks. In this case, they may be contacted again, after the period of time considered acceptable by the treating professional or the research team to invite them to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults living in Buenos Aires with history of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Psychosocial, Cognitive and Health-related Quality Of Life association with symptoms Post COVID-19 syndrome | More than 12 weeks post- acute COVID-19 episode
  Assessment of symptoms and health-related quality of life (ISARIC), fatigue (Chalder fatigue scale and SPHERE questionnaire) and psychosocial evaluation(PHQ-9 and GAD-7 questionnaires)

SECONDARY OUTCOMES:
IL-6, Anti-SARS-Cov-2 S-RBD IgG Antibodies and vitamin D levels | More than 12 weeks post- acute COVID-19 episode
  Evaluate inflammatory, immune and vitamin D profile in post-COVID-19

OTHER OUTCOMES:
Circulating miRNA expression | More than 12 weeks post- acute COVID-19 episode
  RNA-Seq in plasma of participants with persistent symptoms of COVID-19 and comparison

CONTACTS AND LOCATIONS:
Overall Officials: Laura Antonietti, MD, MHA, Principal Investigator — Arturo Jauretche National University; Javier Mariani, MD, Study Chair — Hospital El Cruce; Walter Manucha, PhD, Study Chair — National University of Cuyo; Mariela Paz, PhD, Study Chair — University of Buenos Aires; Martín Rumbo, PhD, Study Chair — Universidad Nacional de La Plata; Liliana Dain, PhD, Study Chair — University of Buenos Aires; Carlos Tajer, Study Chair — Hospital El Cruce
Locations (1):
- Hospital El Cruce, San Juan Bautista, Buenos Aires, Argentina